CLINICAL TRIAL: NCT00760084
Title: An Expanded Access Protocol to Administer Decitabine to Patients With Acute Myelogenous Leukemia or Myelodysplastic Syndrome
Brief Title: Trial of Decitabine in Patients With Acute Myelogenous Leukemia or Myelodysplastic Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Eisai Medical Services, Eisai Inc.
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DACO-021
Record Dates: First submitted 2008-09-24; First posted 2008-09-25 (Estimated); Results first posted 2011-08-02 (Estimated); Last update posted 2011-08-08 (Estimated); Status verified 2011-08

CONDITIONS: Acute Myelogenous Leukemia; Myelodysplastic Syndrome
Keywords: Acute Myelogenous Leukemia; Myelodysplastic Syndrome; Dacogen; Decitabine
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes | interventions — Decitabine

ARMS (1):
- A (Experimental): Decitabine will be administered at a dose of 20 mg/m² over a 1-hour intravenous infusion for 5 consecutive days every 4 weeks.
  Interventions: Drug: Decitabine

INTERVENTIONS:
Drug: Decitabine — Decitabine is administered at a dose of 20 mg/m² over a 1-hour intravenous infusion for 5 consecutive days every 4 weeks in patients with myelodysplastic syndrome (MDS) or acute myeloid leukemia (AML; ≥ 30% blasts).
  Other Names: Dacogen

SUMMARY:
The purpose of this study is to provide decitabine to patients with Acute Myeloid Leukemia (AML) or Myelodysplastic Syndrome (MDS) who have completed participation per protocol in the DACO-018 study.

DETAILED DESCRIPTION:
The objectives of this trial are:

* To generate additional information about the overall safety profile,
* To generate safety information of hepatically or renally impaired patients, as appropriate, and
* To generate safety information when patients are also taking concomitant medications and/or therapies without trial restrictions when decitabine is administered at a dose of 20 mg/m² over a 1-hour intravenous infusion for 5 consecutive days every 4 weeks in patients with MDS or AML (≥ 30% blasts).

The purpose of this open-label, expanded-access trial is to provide decitabine to patients with AML or MDS who have completed participation per protocol in the DACO-018 study and for whom continuation of treatment with decitabine is indicated, per the opinion of the investigator. In order to continue treatment with decitabine, at a minimum, there must be no disease progression while the patient was participating in the DACO-018 trial and during the period after the patient discontinued from the DACO-018 study and before entering this trial. Patients must enroll in this trial within 8 weeks of discontinuing from the DACO-018 study and not have received any other chemotherapy for their disease during this interim period.

Decitabine will be administered at a dose of 20 mg/m² over a 1-hour intravenous infusion for 5 consecutive days every 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Must sign an Institutional Review Board (IRB) -approved informed consent form, indicating his/her awareness of the investigational nature of decitabine and its potential hazards prior to initiation of any study-specific procedures or treatment.
2. Must have had one of the following:

   MDS (de novo or secondary) fitting any of the recognized French-American-British classifications

   OR

   chronic myelomonocytic leukemia (with WBC <12,000/μL)

   AND

   an International Prognostic Scoring System score of ≥1.5 as determined by complete blood count, bone marrow assessment and bone marrow cytogenetics within 30 days of study entry OR AML (≥ 30 % bone marrow blasts), except M3 or acute promyelocytic leukemia.
3. Must be age 18 years or older.
4. Must have completed participation per protocol in the MGI PHARMA DACO-018 decitabine trial.
5. Must enroll in this trial no more than 8 weeks after discontinuation from the MGI PHARMA DACO-018 trial.
6. Must have recovered from all toxic effects of all prior therapy.

Exclusion Criteria:

1. Must not have any other active malignancy, other than basal or squamous cell skin carcinoma.
2. Must not have received in the period after discontinuation from DACO-018 and enrollment into this trial any other chemotherapy agent, including investigational agents, for their disease.
3. Must not have evidence of any other significant clinical disorder or laboratory finding that makes it undesirable for the patient to participate in the trial, at the discretion of the principal investigator.
4. Must not be pregnant or lactating.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2005-07; Primary Completion 2005-09 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Akhil Baranwal, MD, Study Director — Eisai Inc.
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Decitabine: Decitabine will be administered at a dose of 20 mg/m² over a 1-hour intravenous infusion for 5 consecutive days every 4 weeks.
Period: Overall Study
Arm/Group | Decitabine
Started | 10
Completed | 0
Not Completed | 10
Not completed — Physician Decision | 5
Not completed — Withdrawal by Subject | 2
Not completed — Progressive Disease | 3

BASELINE CHARACTERISTICS:
Arm/Group | Decitabine
Number analyzed (Participants) | 10
Age Continuous [Mean (Standard Deviation); unit: years] | 68.5 (11.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 8
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: The Number of Subjects With Adverse Events
Description: Generate safety information when patients were also taking concomitant medications and/or therapies without trial restrictions when decitabine was administered at a dose of 20 milligrams per meter squared (mg/m^2) over a 1-hour intravenous (IV) infusion for 5 consecutive days every 4 weeks in patients with MDS (< 30% blasts) or AML (> 30% blasts).
Time Frame: 3 months
Measure: Number; unit: participants
Arm/Group | Decitabine
Number analyzed (Participants) | 10
participants | 10

ADVERSE EVENTS:
Arm/Group | Decitabine
Serious Adverse Events (participants affected / at risk) | 6/10
Other Adverse Events (participants affected / at risk) | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Decitabine (N=10)
Febrile Neutropenia (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 1
Cardiac Failure Congestive (Cardiac disorders) | 1
Cellulitis Gangrenous (Infections and infestations) | 1
Clostridium Difficile Colitis (Infections and infestations) | 1
Pneumonia Primary Atypical (Infections and infestations) | 1
Pseudomonal Bacteremia (Infections and infestations) | 1
Lung Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Hemorrhage Intracranial (Nervous system disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Decitabine (N=10)
Splenomegaly (Blood and lymphatic system disorders) | 1
Hypothyroidism (Endocrine disorders) | 1
Ocular Hyperaemia (Eye disorders) | 2
Vision Blurred (Eye disorders) | 1
Xerophthalmia (Eye disorders) | 1
Abdominal Pain (Gastrointestinal disorders) | 2
Upper Abdominal Pain (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 3
Diarrhoea (Gastrointestinal disorders) | 3
Gastrointestinal Hemorrhage (Gastrointestinal disorders) | 1
Gingival Bleeding (Gastrointestinal disorders) | 2
Hemorrhoids (Gastrointestinal disorders) | 1
Mouth Hemorrhage (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 4
Proctalgia (Gastrointestinal disorders) | 1
Stomach Discomfort (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
Chest Discomfort (General disorders) | 1
Chest Pain (General disorders) | 2
Chills (General disorders) | 1
Fatigue (General disorders) | 8
Injection Site Reaction (General disorders) | 1
Oedema (General disorders) | 1
Oedema Peripheral (General disorders) | 1
Pain (General disorders) | 2
Pyrexia (General disorders) | 3
Hepatitis (Hepatobiliary disorders) | 1
Perirectal Abscess (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Transfusion Reaction (Injury, poisoning and procedural complications) | 1
Wound (Injury, poisoning and procedural complications) | 1
Blood Uric Acid Increased (Investigations) | 1
Weight Decreased (Investigations) | 2
Glucose Tolerance Impaired (Metabolism and nutrition disorders) | 1
Iron Overload (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Back Pain (Musculoskeletal and connective tissue disorders) | 3
Bone Pain (Musculoskeletal and connective tissue disorders) | 1
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1
Dizziness (Nervous system disorders) | 1
Dysgeusia (Nervous system disorders) | 1
Headache (Nervous system disorders) | 2
Hypoaesthesia (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 2
Insomnia (Psychiatric disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1
Painful Respiration (Respiratory, thoracic and mediastinal disorders) | 1
Paranasal Sinus Hypersecretion (Respiratory, thoracic and mediastinal disorders) | 1
Pleuritic Pain (Respiratory, thoracic and mediastinal disorders) | 1
Respiratiory Tract Infection (Respiratory, thoracic and mediastinal disorders) | 1
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 2
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1
Drug Eruption (Skin and subcutaneous tissue disorders) | 1
Dry Skin (Skin and subcutaneous tissue disorders) | 1
Periorbital Oedema (Skin and subcutaneous tissue disorders) | 1
Petechiae (Skin and subcutaneous tissue disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 1
Rash Generalized (Skin and subcutaneous tissue disorders) | 1
Hot Flush (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No